CLINICAL TRIAL: NCT04255381
Title: Yale-Harvard Hotel-based Closed-Loop Studies in Children (HY-GRAID)
Acronym: HY-GRAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1609018413
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Type1 Diabetes
Keywords: type 1 diabetes; artificial pancreas; closed-loop; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: SIngle arm cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP) (Experimental): Use Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP) system
  Interventions: Device: Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)

INTERVENTIONS:
Device: Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP) — Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)

SUMMARY:
The aim of this clinical study is to determine the feasibility, safety, and preliminary effectiveness of the Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP) system in pediatric subjects with type 1 diabetes in an ambulatory semi-supervised environment over a short duration of 3 days and 2 nights, or up to 60 hours.

DETAILED DESCRIPTION:
The artificial pancreas platform employed under study is centered about the following four key innovations: 1) A zone model predictive control strategy that is at the same time very safe with respect to hypoglycemia, and can simultaneously and independently be tuned with respect to its response to hyperglycemia; 2) Zone control with diurnal blood-glucose target zones; 3) Models of insulin-glucose physiology and insulin on board; 4) A system for alarming and notification of impending hypoglycemia and technical malfunctions: the Health Monitoring System. These features have been evaluated in several clinical trials in adults with unannounced meals and exercise.

The proposed study will evaluate enhancements to our previous system tailored for the special needs of pediatric subjects: 1) A control strategy with responses to hyperglycemia and hypoglycemia spanning wide ranges, as is typical with children; 2) The use of time-dependent zones specific for pediatric subjects; 3) The development of models for young children, capturing the greater physiologic variability, and ensuring cautious insulin delivery; 4) remote alarming and notification systems that are useful to parents.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2- <18 years; for first cohort(s), subjects will be 12-17 years; additional age brackets will be 8-11 years and then <8 years
2. Type 1 diabetes for ≥ 1 year duration - the diagnosis of type 1 diabetes will be based on the history of ketosis/ketoacidosis at diagnosis or laboratory evidence of islet-cell auto-immunity
3. A1c level ≤ 10.0%
4. Use of insulin pump and carbohydrate counting for ≥ 3 months
5. Average total daily insulin dose of at least 10 units/day
6. Current or past use of Continuous Glucose Monitoring (CGM) is desirable but NOT required
7. Normal renal function as measured within 6 months of enrollment
8. Normal thyroid function within 6 months of enrollment, or if previously diagnosed with hypothyroidism, documented within 3 months of enrollment
9. Parent/guardian agrees to stay at hotel with subject for duration of hotel phase and has cell phone that can send/receive text messages
10. Subject and participating parent/guardian speak and comprehend English

Exclusion Criteria:

1. Episode of diabetic ketoacidosis (DKA) within 6 months of enrollment
2. Episode of severe hypoglycemia (seizure, loss of consciousness) within 6 months of enrollment
3. Use of medications (other than insulin) known to affect BG levels within 4 weeks of enrollment - examples include systemic glucocorticoids, metformin, pramlintide, liraglutide)
4. Current use of other medications, that in opinion of investigator, would interfere with safety or effectiveness of the study including acetaminophen
5. Medical disorder, that in opinion of investigator, would be contraindication for inclusion; hypothyroidism and celiac disease are NOT exclusion if under good control
6. Female subjects of childbearing potential unwilling to have pregnancy testing
7. Female subject currently pregnant or lactating
8. History of alcohol or drug abuse, documented eating disorder, or inpatient psychiatric treatment within 6 months of enrollment
9. Subject is currently participating in another research study involving an investigational drug or device

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deshpande S, Weinzimer SA, Gibbons K, Nally LM, Weyman K, Carria L, Zgorski M, Laffel LM, Doyle FJ 3rd, Dassau E. Feasibility and Preliminary Safety of Smartphone-Based Automated Insulin Delivery in Adolescents and Children With Type 1 Diabetes. J Diabetes Sci Technol. 2024 Mar;18(2):363-371. doi: 10.1177/19322968221116384. Epub 2022 Aug 16. PMID 35971681

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 2
  Unknown or Not Reported | 0
Duration of Type I Diabetes [Mean (Standard Deviation); unit: years] | 5.0 (3.2)
Baseline A1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 7.6 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia Safety: Number of Participants With Blood Glucose (BG)) Readings < 50 Milligrams/Deciliter (mg/dL))
Description: Number of participants with more than one confirmed BG < 50 mg/dL
Time Frame: 60 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
Participants
  No more than one confirmed BG < 50 mg/dL | 19
  More than one confirmed BG < 50 mg/dL | 1

2. Primary Outcome: Hyperglycemia Safety: Number of Participants With More Than Two Blood Glucose (BG) Readings > 300 mg/dL Longer Than 2 Hour or Any BG 400 > Milligrams/Deciliter (mg/dL))
Description: No more than two confirmed BG ≥ 300 mg/dL longer than 2 hours, and no BG ≥ 400 mg/dL, unless determined to be from an infusion site failure.
Time Frame: 60 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
Participants
  No more than 2 confirmed BG≥300 mg/dL > 2 hours and no BG≥400 mg/dL not due to infusion site failure | 19
  More than 2 two confirmed BG ≥ 300 mg/dL >2 hours or BG ≥ 400 mg/dL not due to infusion site failure | 1

3. Primary Outcome: Blood Ketone Safety: Number of Participants With Blood Ketone Levels > 1.0 mmol/l for Longer Than 2 Hours or Any Ketone Level> 3.0 mmol/l
Description: Number of participants with blood ketone level > 1.0 mmol/l for longer than 2 hours, and no blood ketone level >3.0 mmol/L, unless determined to be from an infusion site. failure
Time Frame: 60 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
Participants
  blood ketone levels > 1.0 mmol/l for longer than 2 hours | 0
  blood ketone levels > 3.0 mmol/l | 0
  blood ketone levels < 1.0 mmol/l for longer than 2 hours or blood ketone levels < 3.0 mmol/l | 20

4. Primary Outcome: Safety: Number of Participants Who Experienced an Adverse Event
Description: Adverse events include seizure, loss of consciousness, severe hypoglycemia, diabetic ketoacidosis
Time Frame: 60 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
Participants
  seizures | 0
  loss of consciousness | 0
  severe hypoglycemia | 0
  diabetic ketoacidosis | 0
  no adverse event | 20

5. Secondary Outcome: Mean Meter and Sensor Glucose Levels Milligram/Deciliter (mg/dL)
Description: Mean meter and sensor glucose levels (mg/dL)
Time Frame: 60 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
mg/dL
  Meter blood glucose | 161.4 (39.8)
  Sensor glucose | 172 (26)

6. Secondary Outcome: Percent Sensor Glucose Time in Range (70-180 mg/dL)
Description: Percentage of time, over the whole evaluation period, during which the glucose level, as determined by the continuous glucose sensor, is between 70-180 mg/dL
Time Frame: 60 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
percentage of time | 63.5 (14.4)

7. Secondary Outcome: Percent Sensor Glucose Time Below Range (<70 mg/dL)
Description: Percentage of time, over the whole evaluation period, during which the glucose level, as determined by the continuous glucose sensor, is below 70 mg/dL
Time Frame: 60 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
percentage of time | 1.8 (1.4)

8. Secondary Outcome: Percent Sensor Glucose Time Above Range (>180 mg/dL)
Description: Percentage of time, over the whole evaluation period, during which the glucose level, as determined by the continuous glucose sensor, is greater than 180 mg/dL
Time Frame: 60 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
percentage of time | 37.4 (14.8)

9. Secondary Outcome: Percent Sensor Glucose Time in Hypoglycemia (<60 mg/dL)
Description: Percentage of time, over the whole evaluation period, during which the glucose level, as determined by the continuous glucose sensor, is below 60 mg/dL
Time Frame: 60 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
percentage of time | 0.6 (0.7)

10. Secondary Outcome: Percent Sensor Glucose Time in Hyperglycemia (>250 mg/dL)
Description: Percentage of time, over the whole evaluation period, during which the glucose level, as determined by the continuous glucose sensor, is greater than 250 mg/dL
Time Frame: 60 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
percentage of time | 12.1 (10.3)

11. Secondary Outcome: Percent Time AP System Active
Description: Percentage of time, over the whole evaluation period, during which the sensor and pump are determined to be wirelessly connected and communicating with each other, based on duration of alert and error messages indicated by the system
Time Frame: 60 hours
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
Number analyzed (Participants) | 20
percentage of time | 92.7 (7.0)

ADVERSE EVENTS:
Time Frame: 60 hours
Arm/Group | Zone-Model Predictive Control Artificial Pancreas (ZMPC_AP)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04255381/Prot_SAP_000.pdf